CLINICAL TRIAL: NCT06534632
Title: Does Oral Care With Mother's Colostrum Reduce the Risk of Late-Onset Sepsis in Preterm Infants
Brief Title: Oral Care With Colostrum for Preventing Late-onset Sepsis in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Organization for Teaching Hospitals and Institutes (Other)
Responsible Party: Principal Investigator, Marwa Taha, MD, Fellow of Pediatrics (Principal Investigator), General Organization for Teaching Hospitals and Institutes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HM000142
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colostrum group (Experimental): The interventional group received their mother's colostrum through the oropharyngeal route beginning within the first 24 hours of birth and for 5 days at a dose of 0.2 mL/6 hours
  Interventions: Other: Mother's colostrum
- Placebo group (Placebo Comparator): The placebo group received sterile water through the oropharyngeal route beginning in the first 24 hours of birth and for 5 days at a dose of 0.2 mL/6 hours
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Mother's colostrum — Oropharyngeal administration of mother's colostrum
  Arms: Colostrum group
Other: Placebo — Oropharyngeal administration of sterile water
  Arms: Placebo group

SUMMARY:
This clinical trial aimed to evaluate the efficacy of the oral mother's colostrum administration for preventing late-onset sepsis in premature neonates during their stay in the neonatal intensive care unit. The investigators hypothesized that premature infants who receive oral mother's colostrum would have a lower incidence of late-onset sepsis and better hospital outcomes, compared to infants who receive a placebo.

DETAILED DESCRIPTION:
The study was a randomized clinical trial, performed on very-low-birthweight premature newborns admitted to the neonatal intensive care unit of Mataria Teaching Hospital after considering exclusion criteria.

The enrolled newborns were randomly subdivided into two groups (1:1). The colostrum group received their mother's colostrum, and the placebo group received placebo (sterile water) using a standardized protocol. The newborns received 0.2 mL of the colostrum or placebo orally using a swab directed backward into the oropharynx (0.1 mL on either side of the oral cavity), starting during the first 24 hours of life and lasting for 5 days. Vital signs were carefully monitored throughout the procedure. Dosing was provided every 6 hours during the study period.

All infants underwent follow-up from birth until discharge or death whichever came first. Neonates were evaluated for occurrence of late-onset sepsis, death, and other clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Very-low-birth-weight preterm newborns admitted to the neonatal intensive care unit within 24 hours after delivery
* Neonates with gestational age ≤ 34 weeks and weight ≤ 1500 grams

Exclusion Criteria:

* Infants with severe gastrointestinal malformations.
* Infants with serious congenital anomalies or chromosomal abnormalities.
* Infants with signs of early-onset sepsis.
* Any contraindications for breastfeeding because of maternal conditions including active tuberculosis or AIDS, or treatment with medications excreted in breast milk.

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Number of infants with late-onset sepsis in each group | Up to 40 weeks corrected gestational age
  Positive blood cultures collected or clinical symptoms of sepsis after 72 hours of age

SECONDARY OUTCOMES:
Mortality | Up to 40 weeks corrected gestational age
  Number of deaths in each group

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Taha, M.D., Principal Investigator — Mataria Teaching Hospital, General Organization for Teaching Hospitals and Institutes, Egypt; Mai M Mostafa, M.D., Study Director — Mataria Teaching Hospital, General Organization for Teaching Hospitals and Institutes, Egypt; Fifi Helmy, M.D., Study Director — Mataria Teaching Hospital, General Organization for Teaching Hospitals and Institutes, Egypt; Sohaila A Abd El-Halim, M.D., Study Director — Mataria Teaching Hospital, General Organization for Teaching Hospitals and Institutes, Egypt
Locations (1):
- Mataria Teaching Hospital, Cairo, Egypt